CLINICAL TRIAL: NCT05705570
Title: A Phase I Clinical Trial Using Genetically Engineered Autologous T Cells to Express Chimeric Antigen Receptor (CAR) for Treatment of Patients With Refractory or Relapsed CD19-positive B Lymphoid Malignancies
Brief Title: Clinical Trial Using CAR- T Cells for Treatment of Patients With Refractory or Relapsed CD19-positive B Lymphoid Malignancies
Acronym: CARTHIAE-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nelson Hamerschlak (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nelson Hamerschlak, MD, PhH, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30173220.5.0000.0071
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia Refractory; B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory; Chronic Lymphocytic Leukemia Recurrent; Chronic Lymphocytic Leukemia Refractory
Keywords: CAR T cell; CD19+ B-cell Malignancies
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: A phase I study, with a "3+3" dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide + Fludarabine + Infusion of CAR-T Cells (Experimental): Lymphodepleting regimen, consisting of Cyclophosphamide 60mg/kg IV on day -6 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of Chimeric antigen receptor T-cells (CAR-T) on day 0
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Chimeric antigen receptor T cells to be implemented in a "3 + 3" design on day 0

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60mg/Kg on day -6
Drug: Fludarabine — Fludarabine 25mg/m^2 IV on days -5 to -3
Biological: Chimeric antigen receptor T cells to be implemented in a "3 + 3" design on day 0 — Level -1 (1 x 105 cells/kg)
  Level 1 [Starting dose] (5 x 105 cells/kg)
  Level 2 (1 x 106 cells/kg)
  Level 3 (2 x 106 cells/kg)

SUMMARY:
This is a phase l, single arm, prospective open, dose-escalation study in patients with relapsed or refractory CD19-positive B cell malignancies (ALL, NHL, CLL). The trial will include adult and pediatric patients. There will be three individual cohorts, defined by disease biology: pediatric ALL and aggressive pediatric NHL (Cohort 1), adult ALL (Cohort 2) and adult NHL/CLL (Cohort 3).

DETAILED DESCRIPTION:
The investigators will evaluate the safety of the MB-CART19.1 and determine the recommended dose levels for the Phase II clinical trial.

Dose evaluation will start in Cohorts 1 and 2 with Dose Level 1 (5x10e5 CAR T cells/Kg) and in Cohort 3 with Dose Level 2 1x10e6 CAR T cells/Kg) , sparing Dose Level 1 . Each of the cohorts will evaluate the safety of the CAR-T cells.

In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD. In Dose Level 3, three additional patients will be treated, if no DLT occurred. Dose Level 0 will be tested only if Dose Level 1 is not tolerable.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have relapsed or refractory ALL, lymphoma or CLL treated with at least two lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve partial or complete remission with the last regimen.

   Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) subjects are eligible if they progressed, had stable disease or relapsed after two lines of therapy, including tyrosine kinase inhibitors (TKIs).

   Subjects with DLBCL must have progressed, had SD, or recurred after initial treatment regimens that include an anthracycline and an anti-CD20 monoclonal antibody.

   Subjects with transformed FL, MZL, or CLL/SLL must have progressed, had SD or recurred with transformed disease after initial treatment for DLBCL.

   Subjects who relapse ≥12 months after therapy should have progressed after autologous transplant or been ineligible for autologous transplant.
2. 2. The patient's disease must be CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available.
3. Age 2 to 70 years.
4. Performance status: Adult Subjects: ECOG ≤ 2 for patients ≥ 16 years; Subjects < 16 years of age: lansky ≥ 50%
5. Normal Organ and Marrow Functioning (supportive treatment is allowed according to institutional standards, i.e. filgrastim, transfusion)

   • Total Bilirubin ≤ 2; AST (SGOT) ≤ 5 times the upper limit of normal; ALT (SGTP) ≤ 5 times the upper limit of normal; Serum creatinine ≤ 1.5; Pulse oximetry >91% on room air; No dyspnea or mild dyspnea (≤ Grade 1); Forced expiratory volume in 1 s (FEV1) ≥50% or carbon monoxide diffusion test (DLCO) ≥50% of predicted level; Left ventricular ejection fraction ≥ 45% confirmed by echocardiogram; Subjects must have the following hematologic function parameters: Neutrophils > 1000/uL; Absolute Lymphocyte Count > 100/uL; Platelets ≥ 50,000/L Patient should not be excluded if change of the above parameters due to spinal cord disease infiltration;
6. Prior therapy wash-out - At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives, Blinatumomab with 4 months prior CAR-T infusion.
7. For women of reproductive potential: use a highly effective contraceptive for at least 1 month prior to screening and agree to use a method during study participation and for an additional 4 months after CAR T-cell administration has ended.
8. Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Autologous transplant within 6 weeks of planned CAR-T cell infusion;
2. History of allogeneic stem cell transplant 4 months prior CAR T cell infusion.
3. Use of immunosuppression therapy;

   • Patients must have completed immunosuppression therapy; Systemic corticosteroid therapy must be stopped more than 72 hours after infusion; Systemic drugs for graft-versus-host disease should be withheld at least 4 weeks prior to infusion;
4. Presence of graft-versus-host disease Grade ≥ 2;
5. Receiving CAR T cell treatment outside of this protocol;
6. Active central nervous system or meningeal involvement by tumor. Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast-enhanced MRI imaging for at least 90 days prior to registration.
7. History of active malignancy other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast).
8. HIV infection; HTLV
9. Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
10. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects.
11. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
12. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
13. Serious and/or potentially fatal medical conditions
14. Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
15. History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.
16. Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation, e.g. as part of the mandatory lymphodepletion protocol, pre-medication for infusion, rescue medication/salvage therapies for treatment related toxicities;

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the recommended dose of CAR-T cells for a future phase II study | Until day 28 after CAR-T cells infusion
  The RP2D will be the maximum tolerated dose (MTD) or the highest dose studied if an MTD is not obtained.

SECONDARY OUTCOMES:
Response to treatment for each timepoint. | day 28
  ORR in ALL (Rate of CR/CRh)
Response to treatment for each timepoint | day 28, patients not in CR on day 28: month 3
  ORR in NHL/CLL (Rate of CR/CRh)
Assess overall survival (OS), progression-free survival (PFS). | at 1 year after CAR-T infusion
  Overall survival (OS) and progression-free survival (PFS) will be assessed by dose cohort and in the first two groups at the MTD (or at the highest dose studied).
Phenotype and persistence of CAR-T | days 2, 7, 10, 14, 28, weeks 8, 12, months 6, 12, 24, 36, 48, 60
  Blood samples for determination of persistence/phenotyping of infused CAR-T cells will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Hamerschlak, MD, PhH, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No